CLINICAL TRIAL: NCT00004650
Title: Phase III Randomized Study of the Effect of Postmenopausal Estrogen Replacement Therapy on Alveolar Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Collaborators: Washington University School of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11726; WUSM-900449
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: Osteoporosis
Keywords: disease-related problem/condition; osteoporosis; rare disease
MeSH Terms: conditions — Osteoporosis; Rare Diseases | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone

INTERVENTIONS:
Drug: conjugated estrogens
Drug: Medroxyprogesterone

SUMMARY:
OBJECTIVES: I. Quantify periodontal alveolar bone loss rates in postmenopausal women.

II. Evaluate the effects of estrogen on alveolar bone loss rates in these patients.

III. Determine whether changes in periodontal bone mass relate to bone mass changes in other skeletal sites in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind, placebo controlled study. Patients are randomly assigned to receive placebo or conjugated estrogens and, if no prior hysterectomy, medroxyprogesterone. Patients also receive calcium supplementation therapy daily for 3 years.

Participants in the placebo group may be removed from study if bone loss exceeds 5% per year.

A study duration of 3 years is anticipated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Women postmenopausal for at least 2 years
* At least 10 teeth for which radiographic measurements can be obtained, i.e.: Not severely tilted Not so closely spaced that interproximal bone is thin Not in positions of restricted access

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1993-08

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Hildebolt, Study Chair — Washington University School of Medicine

REFERENCES:
- [Background] Hildebolt CF, Pilgram TK, Dotson M, Yokoyama-Crothers N, Muckerman J, Hauser J, Cohen S, Kardaris E, Vannier MW, Hanes P, Shrout MK, Civitelli R. Attachment loss with postmenopausal age and smoking. J Periodontal Res. 1997 Oct;32(7):619-25. doi: 10.1111/j.1600-0765.1997.tb00940.x. PMID 9401935
- [Background] Hildebolt CF. Osteoporosis and oral bone loss. Dentomaxillofac Radiol. 1997 Jan;26(1):3-15. doi: 10.1038/sj.dmfr.4600226. PMID 9446984
- [Background] Hildebolt CF, Brunsden B, Yokoyama-Crothers N, Pilgram TK, Townsend KE, Vannier MW, Shrout MK. Comparison of reliability of manual and computer-intensive methods for radiodensity measures of alveolar bone loss. Dentomaxillofac Radiol. 1998 Jul;27(4):245-50. doi: 10.1038/sj/dmfr/4600352. PMID 9780904